CLINICAL TRIAL: NCT04249050
Title: Effects of Immunonutrition on the Acute Immune Response in Hospitalized Patients With Pneumonia
Brief Title: Effects of Immunonutrition in Patients With Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-19088763
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Pneumonia; Lung Infection; Muscle Loss; Malnutrition; Pulmonary Disease
MeSH Terms: conditions — Pneumonia; Muscular Atrophy; Malnutrition; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group is receiving a nutritional drink containing potential immune stimulating ingredients (fish oil, arginine, nucleotides)
  Interventions: Dietary Supplement: Oral Impact powder
- Control group (No Intervention): The Control group is receiving the hospital´s Standard Of Care.

INTERVENTIONS:
Dietary Supplement: Oral Impact powder — Oral nutritional supplement containing fish oil, arginine and RNA
  Arms: Intervention group

SUMMARY:
The project is a randomized controlled trial taking place in the North Zealand hospital in the city Hilleroed, Denmark.

The aim is to investigate the potential beneficial effects of immunonutrition containing fish oil, arginine and RNA, on the acute immune response in patients with pneumonia.

DETAILED DESCRIPTION:
Immunonutrition has a well-documented beneficial effect on surgical patients by strengthening the immune system and reducing the following: inflammation, the number of infections as well as hospitalization time. A study in operated patients demonstrated the benefit of immunonutrition by reducing unwanted inflammation, measured by the pro-inflammatory signalling protein, interleukin-6. The same study saw a smaller decrease in immune function (measured as the level of phagocytosis) in the group receiving immunonutrition than in the control group. This project will investigate whether similar effects can be detected in patients with pneumonia.

The project is being carried out in a collaboration between the University of Copenhagen, The main hospital of Copenhagen (Rigshospitalet) and North Zealand Hospital. The project is a randomized clinical intervention study, which spans 10 days. Participants are allocated to the intervention group or the control group. The project is being carried out at the North Zealand hospital, at the Department of Pulmonary- and Infectious Diseases.

The intervention group receives the department's standard treatment (Standard Of Care) + immunonutrition, while the control group receives the hospital department's standard treatment (Standard Of Care). On a daily basis, the patient's clinical condition and the activity of the immune system is measured for the purpose of determine whether there is an effect of immunonutrition.

ELIGIBILITY:
Inclusion Criteria:

* Authorized individuals diagnosed with pneumonia who speak and write in danish

Exclusion Criteria:

* individuals with Immunodeficiency
* individuals with another primary diagnose
* individuals with an allergy against product ingredients
* individuals with dementia
* individuals with dysphagia
* individuals with cancer in treatment
* individuals with Chronic Obstructive Pulmonary Disease on continuing steroid treatment or home administered oxygen treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Interleukin-6 | daily measure from first day of inclusion until discharge (maximum 10 days)
  Measure of the acute immune response

SECONDARY OUTCOMES:
Length of stay | From admittance to discharge (maximum 10 days)
  Measure of hospitalized days
Hand grip strength | Daily from admittance to discharge (maximum 10 days)
  Measure of the mobilization of strength

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte L Madsen, M.D., Ph.D., Principal Investigator — North Zealand Hospital, Hilleroed, Denmark
Locations (1):
- Department of Lung Medicine and Infectious Diseases, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Braga M, Gianotti L, Vignali A, Carlo VD. Preoperative oral arginine and n-3 fatty acid supplementation improves the immunometabolic host response and outcome after colorectal resection for cancer. Surgery. 2002 Nov;132(5):805-14. doi: 10.1067/msy.2002.128350. PMID 12464864
- [Result] Marimuthu K, Varadhan KK, Ljungqvist O, Lobo DN. A meta-analysis of the effect of combinations of immune modulating nutrients on outcome in patients undergoing major open gastrointestinal surgery. Ann Surg. 2012 Jun;255(6):1060-8. doi: 10.1097/SLA.0b013e318252edf8. PMID 22549749